CLINICAL TRIAL: NCT05817175
Title: International Prospective REgistry on Pre-pectorAl Breast REconstruction
Acronym: I-PREPARE
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: EUBREAST ETS (Unknown)
Responsible Party: Principal Investigator, Oreste Davide Gentilini, Professor, Head of Breast Surgery Unit, IRCCS San Raffaele
Other Study IDs: EUBREAST-11R
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast reconstruction; Pre-pectoral Breast Prosthesis; Mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pre-pectoral breast reconstruction — to prospectively evaluate the utilization of the pre-pectoral approach, and evaluate oncological and aesthetic outcomes related to each type of surgical technique and the use of postmastectomy radiation therapy

SUMMARY:
This is an international multicenter prospective cohort study aimed at collecting data on breast reconstruction techniques with pre-pectoral implants after mastectomy for breast cancer. The aim of the study is to collect data on the surgical, aesthetic and oncological results, as well as on the quality of life of the patients who will undergo breast reconstruction with a pre-pectoral approach.

DETAILED DESCRIPTION:
1,236 patients undergoing mastectomy for breast cancer and subsequent pre-pectoral breast reconstruction will be enrolled. Being an observational study, the diagnostic-therapeutic path of the patients will not be modified in any way. Therefore, no risks are anticipated for the patients who will participate in this study. Potential benefits deriving from the study will be for future patients for whom good quality data will be available which can guide the choice of the type of breast reconstruction to be performed, in particular the most appropriate type of technique in the pre-pectoral approach.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 18 years old
* Signed informed consent form
* Patients undergoing mono or bilateral therapeutic mastectomy
* Patients undergoing pre-pectoral implant-based breast reconstruction with implant or expander with or without mesh

Exclusion Criteria:

* Male patients
* Patients not suitable for surgical treatment
* Patients undergoing subpectoral reconstruction
* Patients undergoing breast reconstruction with autologous tissue.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients older than 18 years old
Study Population: All patients who are candidates for implant-based reconstruction should be informed about the possible participation to this clinical study. The inclusion and exclusion criteria are verified by the investigator and an informed consent is obtained from the patient.
  The therapeutic pattern should be followed according to institutional and national standards. Since this is a non-interventional trial, the study sites do not deviate from their own study protocol at any timepoint.
Sampling Method: Non-Probability Sample
Enrollment: 1236 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Implant-loss at three months postoperatively | three months postoperatively
  Rate of implant-loss at three months postoperatively defined as the unplanned removal or loss of the implant as a result of infection or other complication

SECONDARY OUTCOMES:
Number of patients with Infection | three months postoperatively
  Rate of infection defined as minor if oral antibiotic was required, major if surgical revision and/or hospitalisation was necessary;
Number of patients with re-admission and re-operation | three months postoperatively
  Rate of re-admission and re-operation
Evaluation of Quality of life | 0, 6, 12 and 24 months
  Patient's satisfaction and quaity of life measured through BREASTQ (Breast Reconstruction Module Questionnaire)
Number of Early onset complication | three months postoperatively
  Early onset complication at 3 month follow up: seroma, hematoma/bleeding, skin flap or T junction necrosis, nipple necrosis, wound dehiscence, implant malposition (i.e. rotation, displacement etc..), red-breast syndrome
Number of late-onset complications | 6-12-24 months
  seroma, capsular contracture, wrinkling/rippling, implant malposition (i.e. rotation, displacement etc..) implant upper pole visibility, implant loss;

CONTACTS AND LOCATIONS:
Overall Officials: Oreste D Gentilini, Dr, Study Chair — IRCCS San Raffaele
Locations (11):
- Univesidad de Buenos Aires, Buenos Aires, Argentina
- Egypt (2):
  - Mansoura Insurance, Al Mansurah
  - Mansoura Oncology, Al Mansurah
- National ans Kapodistrian University of Athens, Athens, Greece
- Italy (2):
  - Ospedale San Raffaele, Milan, MI
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma, RM
- University Hospital of Karol Marcinkowski, Zielona Góra, Poland
- Prof. Dr. Ion Chiricuta Institute of Oncology, Cluj-Napoca, Romania
- Hospital del Mar, Barcelona, Spain
- Marmara University School of medicine, Istanbul, Turkey (Türkiye)
- University Hospitals of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No